CLINICAL TRIAL: NCT00047658
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Biology, and Clinical Effects of Interferon Gamma-1b Administered Subcutaneously to Patients With IPF Followed by an Open-Label Extension
Brief Title: A Study of the Safety and Clinical Effects of Interferon Gamma-1b in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InterMune (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIPF-002
Record Dates: First submitted 2002-10-09; First posted 2002-10-11 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Interferon-gamma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Interferon-gamma 1b — 200 mcg, SQ, 3x per week

SUMMARY:
Study GIPF-002 is a phase 2 study designed to characterize the biologic and clinical effects of IFN-g 1b. The objective of the Study is to characterize the biologic and clinical effects of IFN-g 1b administered to patients with idiopathic pulmonary fibrosis (IPF). The Study will be conducted at multiple sites and enroll 30 patients with IPF who have failed treatment with corticosteroids.

ELIGIBILITY:
Male or Female 20-79 years old

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2001-11; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
change in percent predicted FVC, resting arterial blood gas assessment of alveolar-arterial oxygen gradient, percent predicted DLCO, dyspnea scale, baseline dyspnea index/transition dyspnea index | 23 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Williamson Bradford, MD, Study Director — InterMune
Locations (1):
- UCLA, Dept. of Medicine, Los Angeles, California, United States